CLINICAL TRIAL: NCT04511728
Title: A Multi-center, Randomized, Single-blind, Propofol Injectable Emulsion Parallel-controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of HSK3486 Injectable Emulsion in the Induction of General Anesthesia in Patients Undergoing Elective Surgery
Brief Title: A Study to Evaluate the Efficacy and Safety of HSK3486 in the Induction of General Anesthesia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSK3486-306
Record Dates: First submitted 2020-08-11; First posted 2020-08-13 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Induction and Maintenance of General Anesthesia
MeSH Terms: interventions — HSK3486; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HSK3486 (Experimental)
  Interventions: Drug: HSK3486
- Propofol (Active Comparator)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: HSK3486 — The initial Induction dose of HSK3486 is 0.4 mg/kg. The initial maintenance dose of HSK3486 is 0.8 mg/kg/h
  Arms: HSK3486
Drug: Propofol — The initial Induction dose of propofol is 2.0 mg/kg. The initial maintenance dose of propofol is 5.0 mg/kg/h
  Arms: Propofol

SUMMARY:
This is a multi-center, randomized, single-blind, propofol injectable emulsion parallel-controlled Phase III clinical study. A total of patients undergoing elective surgery are intended to be enrolled and randomly assigned to HSK3486 group and propofol group in a 2:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. In-patients undergoing non-emergency, non-cardiothoracic, and non-extracerebral elective surgeries with expected operation time ≥ 1 h and requiring tracheal intubation under general anesthesia (patients whose surgery type may affect the collection of BIS parameter should not be included);
2. Male or female, age ≥ 18 and ≤ 65 years old;
3. American Society of Anesthesiologists (ASA) class I-III;
4. Body mass index (BMI) ≥ 18 and ≤ 30 kg/m^2;
5. Vital signs in the screening period meeting the following criteria:

   1. Respiration rate ≥ 10 and ≤ 24 breaths/min;
   2. SpO2 while breathing ≥ 95%;
   3. Systolic blood pressure ≥ 90 mmHg and ≤ 160 mmHg;
   4. Diastolic blood pressure ≥ 60 mmHg and ≤ 100 mmHg;
   5. Heart rate ≥ 55 and ≤ 100 bpm. (Note: The heart rate is judged by the results of ECG monitoring after signing the ICF, and the heart rate results of 12-lead ECG examination are not used as the basis for judgment.)
6. Subjects must understand the procedures and methods of this study, and be willing to provide informed consent and to complete the trial in strict accordance with study protocol.

Exclusion Criteria:

1. Patients with contraindications to general anesthesia or previous history of anesthesia accidents;
2. Known hypersensitivity to excipients and ingredients found in propofol injection and HSK3486 injectable emulsion (soybean oil, glycerin, triglycerides, egg lecithin, sodium oleate, and sodium hydroxide), benzodiazepines, opioids, rocuronium bromide, and sugammadex sodium; cross-reactivity to halogenated anesthetics, jaundice or unexplained fever from previous use of halogenated anesthetics; contraindications to propofol;
3. The following disease history or evidence that increases the risk of sedation/anesthesia is collected before/during screening:

   1. History of cardiovascular diseases: uncontrolled hypertension or SBP > 160 mmHg and/or DBP > 100 mmHg after treatment with antihypertensive drugs, severe arrhythmia, heart failure, Adams-Stokes syndrome, unstable angina, myocardial infarction, tachycardia/bradycardia requiring medication, or third-degree atrioventricular block within 6 months before screening, or QTcF interval of ≥ 450 ms (corrected using Fridricia's formula) during the screening period;
   2. History of respiratory diseases: respiratory insufficiency, history of obstructive pulmonary disorders, history of bronchospasm requiring treatment within 3 months before screening, and acute respiratory infection with one of the symptoms such as obvious fever, wheezing or productive cough within 1 week before the baseline period;
   3. History of neurological and psychiatric disorders: craniocerebral injury, convulsions, epilepsy, intracranial hypertension, cerebral aneurysms, cerebrovascular accidents; or schizophrenia, mania, long-term use of psychotropic drugs, history of cognitive impairment, etc.;
   4. History of gastrointestinal tract diseases: gastrointestinal retention, active bleeding, gastroesophageal reflux or obstruction, etc. which may cause reflux and aspiration judged by the investigator;
   5. Diabetic patients with uncontrolled blood glucose (fasting blood glucose ≥ 11.1 mmol/L, and/or random blood glucose ≥ 13.6 mmol/L);
   6. Patient with a history of uncontrolled and clinically significant liver, kidney, blood system, nervous system or metabolic system diseases judged by the investigator to be unsuitable for this trial;
   7. History of alcohol abuse within 3 months prior to screening, where alcohol abuse refers to daily alcohol drinking > 2 units of alcohol (1 unit = 360 mL of beer or 45 mL of liquor with 40% alcohol or 150 mL of wine);
   8. History of drug abuse within 3 months prior to screening;
   9. Serious infection, trauma, or major surgery within 4 weeks prior to screening.
4. Any of the following respiratory management risks before/during screening:

   1. Asthma history and stridor;
   2. Sleep apnea syndrome;
   3. History or family history of malignant hyperthermia;
   4. History of intubation failure;
   5. Judged by the investigator to have difficult airway or judged as difficult tracheal intubation (modified Mallampati score III or IV).
5. In receipt of any of the following drugs or therapies prior to screening:

   1. Participated in other clinical drug trials within 1 month prior to screening;
   2. Used drugs that may affect QT intervals within 2 weeks prior to screening;
   3. In receipt of propofol, other general sedatives/anesthetics, and/or opioid analgesics or compounds containing opioid analgesics within 3 days prior to screening.
6. Patient whose laboratory test results measured at screening reach the following criteria and are verified through re-examination:

   1. Neutrophil count ≤ 1.5 × 10^9/L;
   2. Platelet count < 80 × 10^9/L;
   3. Hemoglobin < 90 g/L (no blood transfusion within the last 14 days);
   4. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 3.0 × ULN;
   5. Total bilirubin > 2 × ULN;
   6. Blood creatinine > 1.5 × ULN.
7. Women who are pregnant or breastfeeding; women of child-bearing potential or men who are unwilling to use contraception method during the trial; subjects who are planning pregnancy within 3 months after the completion of the trial (including male subjects);
8. Subjects judged by the investigator to be unsuitable for participating in this trial for any reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Success rate of anesthesia maintenance | During maintenance of general anesthesia on day 1
  During the maintenance of anesthesia, the subject is not recovered and no remedial anesthetic is used

SECONDARY OUTCOMES:
Success rate of anesthesia induction | During induction of general anesthesia on day 1
  During the induction of anesthesia, the subject achieves successful induction (i.e., MOAA/S ≤ 1) after administration of the study drug (up to 2 top-up doses), and no remedial anesthetic is used.
Percentage of time from the beginning of surgical skin incision to the end of surgery | During maintenance of general anesthesia on day 1
  when bispectral index (BIS) is ≥ 40 and ≤ 60.
Time to recovery from anesthesia | A period of time from discontinuation of the study drug to recovery after the end of surgery on day 1
  3 consecutive MOAA/S = 5. Record the time when MOAA/S = 5 is reached for the first time.
Time to respiratory recovery | A period of time from discontinuation of the study drug to respiratory recovery after the end of surgery on day 1
  Respiratory rate ≥ 8 breaths/min and the tidal volume ≥ 5 mL/kg
Time from discontinuation of the study drug to 3 consecutive Aldrete score ≥ 9. | A period of time from discontinuation of the study drug to 3 consecutive Aldrete score ≥ 9 on day 1
Number of patients with adverse events | Pre-dose to 48 hours post-dose
  Safety endpoints

OTHER OUTCOMES:
Concentrations of HSK3486 and propofol in blood samples (sporadic sampling). | The end of the induction administration (to start of the maintenance administration) to 1~6 hours post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital，Sichuan University, Chengdu, China

REFERENCES:
- [Derived] Liang P, Dai M, Wang X, Wang D, Yang M, Lin X, Zou X, Jiang K, Li Y, Wang L, Shangguan W, Ren J, He H. Efficacy and safety of ciprofol vs. propofol for the induction and maintenance of general anaesthesia: A multicentre, single-blind, randomised, parallel-group, phase 3 clinical trial. Eur J Anaesthesiol. 2023 Jun 1;40(6):399-406. doi: 10.1097/EJA.0000000000001799. Epub 2023 Jan 19. PMID 36647565